CLINICAL TRIAL: NCT00586196
Title: Supporting the Health of Adults Undergoing Orthopedic Surgery During the Recovery Period
Acronym: SHARP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Edward Marcantonio, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2006p-000193; R21AG027549 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Delirium
Keywords: Delirium; Postoperative confusion; Hip fracture; Long bone fracture
MeSH Terms: conditions — Delirium; Hip Fractures | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: donepezil
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil — 5 mg each day for 30 days
  Other Names: Aricept
  Arms: 1
Drug: Placebo — Encapsulated cornstarch One capsule daily for 30 days
  Arms: 2

SUMMARY:
Delirium (acute confusion) is a highly prevalent condition among hospitalized elders with substantial morbidity within the hospital and beyond. Particular patient populations are at high risk for poor outcomes after an episode of delirium. Patients with hip and other long bone fractures are at increased risk of developing delirium (acute confusion) which impedes functional recovery. This is a pilot study to test the tolerability and efficacy of donepezil, a cholinesterase inhibitor medication used commonly in persons with dementia, for the prevention of new or worsening delirium in aged hip and other long-bone fracture patients. Additional purposes involve gathering a small amount of patients' serum to better understand the pathophysiology of delirium in this population.

The purposes of this pilot study are to determine: 1) the safety and tolerability a cholinesterase inhibitor medication) in aged hip and long bone fracture patients, 2) To obtain estimates of subject accrual and preliminary estimates of effect size on the development of new delirium symptoms to allow for planning of a larger, definitive trial, 3) To better understand the underlying causes of delirium by examining whether a measure of blood anticholinergic activity relates to the incidence and persistence of delirium symptoms, and 4) To explore the interaction between anticholinergic activity, donepezil therapy, and delirium symptoms.

ELIGIBILITY:
Inclusion Criteria:

* hip or other long bone fracture undergoing operative repair
* age of 70 years or older
* the ability to communicate effectively in English (including adequate hearing)
* residence within a 50 mile radius of the BIDMC
* life expectancy 6 months or greater
* not currently on cholinesterase inhibitor therapy
* not with known hypersensitivity to cholinesterase inhibitors
* not a previous study participant or refusal

Exclusion Criteria:

* patients with sick sinus syndrome or greater than 1st degree AV block without a pacemaker
* patients with a pathologic fracture due to metastatic cancer
* patients with advanced dementia or total functional dependence.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Marcantonio, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Marcantonio ER, Palihnich K, Appleton P, Davis RB. Pilot randomized trial of donepezil hydrochloride for delirium after hip fracture. J Am Geriatr Soc. 2011 Nov;59 Suppl 2(Suppl 2):S282-8. doi: 10.1111/j.1532-5415.2011.03691.x. PMID 22091574

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil : 5 mg Each Day for 30 Days: donepezil : 5 mg each day for 30 days
- Placebo : Encapsulated Cornstarch: Placebo : Encapsulated cornstarch One capsule daily for 30 days
Period: Overall Study
Arm/Group | Donepezil : 5 mg Each Day for 30 Days | Placebo : Encapsulated Cornstarch
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil : 5 mg Each Day for 30 Days | Placebo : Encapsulated Cornstarch | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 88 (5.2) | 87 (3.7) | 87 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Delirium Using the CAM Over Time
Description: Confusion Assessment Method (CAM)-Measure of the presence or absence of delirium. Requires 1) acute change with fluctuating course, 2) inattention, and either 3) disorganized thinking or 4) altered level of consciousness.
Time Frame: Baseline, hospital interviews, weeks 2, 4 and 6
Measure: Number; unit: percentage of participants
Arm/Group | Donepezil : 5 mg Each Day for 30 Days | Placebo : Encapsulated Cornstarch
Number analyzed (Participants) | 7 | 9
percentage of participants
  basline | 14 | 44
  hospital interviews | 64 | 64
  Week 2 | 43 | 43
  week 4 | 17 | 43
  week 6 | 50 | 50
Statistical Analysis 1: Comparison: Donepezil : 5 mg Each Day for 30 Days vs Placebo : Encapsulated Cornstarch; Test type: Superiority or Other; GEE; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 2.3]

2. Secondary Outcome: Change From Baseline and MDAS Scores Over Time
Description: Measures severity of 10 delirium symptoms items (0 not present, 1 mild, 2 moderate, 3 severe) yielding a total score of 0 to 30, with 30 most severe.
Time Frame: Baseline, hospital discharge, weeks 2, 4 and 6
Population: Based on ability to recruit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil : 5 mg Each Day for 30 Days | Placebo : Encapsulated Cornstarch
Number analyzed (Participants) | 7 | 9
units on a scale
  Baseline | 6.3 (3.4) | 8.4 (6.5)
  Change at Hospital Discharge | 1.3 (2.5) | 1.6 (5.2)
  Change at Week 2 | -0.1 (2.3) | -2.2 (4.9)
  Change at week 4 | -1.2 (3.5) | -2.0 (6.4)
  Change at week 6 | -0.6 (2.6) | -2.0 (7.5)
Statistical Analysis 1: Comparison: Donepezil : 5 mg Each Day for 30 Days vs Placebo : Encapsulated Cornstarch; Test type: Superiority or Other; GEE; Effect Size = -0.2, 95% CI 2-sided [-1.5 to 1.2]

ADVERSE EVENTS:
Arm/Group | Donepezil : 5 mg Each Day for 30 Days | Placebo : Encapsulated Cornstarch
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/9
Other Adverse Events (participants affected / at risk) | 7/7 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil : 5 mg Each Day for 30 Days (N=7) | Placebo : Encapsulated Cornstarch (N=9)
Serious Adverse Event (General disorders) | 2 (2) | 0 (0) — Serious adverse events were collected non-specifically and all were deemed unlikely to study participation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil : 5 mg Each Day for 30 Days (N=7) | Placebo : Encapsulated Cornstarch (N=9)
Insomnia (Nervous system disorders) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1
Frequency of Urination (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes